CLINICAL TRIAL: NCT03560726
Title: Telehealth Cognitive Behavioral Stress Management for Adults With Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Responsible Party: Principal Investigator, Christina Bathgate, Licensed Clinical Psychologist, National Jewish Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3143
Record Dates: First submitted 2018-05-03; First posted 2018-06-18 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Anxiety; Depression; Stress; Coping Skills; Cystic Fibrosis
MeSH Terms: conditions — Anxiety Disorders; Depression; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth (Experimental): Participants randomized into the telehealth arm will receive up to 7 one-hour telehealth visits with the study psychologist. The first six sessions will focus on cognitive behavioral stress management topics and the seventh session is optional, focusing on lung transplant readiness. Participants will fill out questionnaires every other week (baseline, week 2, week 4, week 6, week 8) and during a 3-month follow-up (week 20). Participants will wear an actigraphy watch to track sleep and movement for one week at a time during baseline, week 8, and week 20.
  Interventions: Behavioral: Cognitive Behavioral Stress Management
- Treatment-As-Usual (TAU) (No Intervention): Participants randomized into the TAU arm will not receive any telehealth visits during the 8-week intervention phase. Participants will fill out questionnaires every other week (baseline, week 2, week 4, week 6, week 8) and during a 3-month follow-up (week 20).
  Participants will wear an actigraphy watch to track sleep and movement for one week at a time during baseline, week 8, and week 20.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Stress Management — Cognitive behavioral stress management is a well-established, practical intervention that combines elements of cognitive behavioral therapy with techniques designed to improve coping skills, social support, communication, and relaxation/mindfulness.
  Arms: Telehealth

SUMMARY:
The purpose of this study to to assess the feasibility, acceptability, and satisfaction of a telehealth cognitive behavioral stress management (CBSM) intervention among adults with cystic fibrosis (CF) who exhibit elevated anxiety and/or depression symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Fluent in English
* Diagnosed with Cystic Fibrosis
* Colorado resident
* Access to personal device (smart phone, computer, tablet) with 1) reliable internet connection, and 2) a built-in web camera and microphone or the capability to install a study-provided web camera and microphone
* Regular access to a private location with sufficient lighting that is free from distractions or intrusions to use during telehealth sessions
* Access to private email to complete surveys
* Mild anxiety and/or depression symptoms (i.e., a score of 5 or higher on the Generalized Anxiety Disorder 7 Item Scale (GAD-7) and/or the Patient Health Questionnaire 9 Item Scale (PHQ-9))

Exclusion Criteria:

* Currently receiving therapy or counseling with an outside provider for a mental health condition
* Currently in treatment for alcohol or substance abuse
* Unstable medical condition (not including cystic fibrosis)
* Neurological disease
* Pregnant women
* Active suicidal intent or plan (a score of 1 or higher on the Suicide Severity Scale)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Feasibility (patient perspective) | Week 0 (baseline)
  Assess the feasibility of telehealth-delivered Cognitive Behavioral Stress Management from the patient perspective using participation rates (i.e., number of people interested and consented into the study).
Feasibility (clinician perspective) | Week 8
  Assess the feasibility of telehealth-delivered Cognitive Behavioral Stress Management from the clinician perspective using the Structured Assessment of Feasibility (SAFE; 16 items). The first 8 items provide information about barriers to implementation and the second 8 items provide information about enablers to implementation. It is recommended that no overall summary score be used, as this scale is designed to highlight barriers and facilitators that future programs should consider if they decide to continue or begin implementing this intervention.
Acceptability (patient perspective 1 of 2) | Week 8
  Assess the acceptability of telehealth-delivered Cognitive Behavioral Stress Management from the patient perspective using participation rates (i.e., telehealth sessions completed, dropouts).
Acceptability (patient perspective 2 of 2) | Week 8
  Assess the acceptability of telehealth-delivered Cognitive Behavioral Stress Management from the patient perspective using the Acceptability Scale (12 items; 5 = strongly agree, 1 = strongly disagree), which was adapted specifically for this study. A mean acceptability score will be computed from these 12 items.
Satisfaction (patient perspective 1 of 2) | Week 8
  Assess the satisfaction of telehealth-delivered Cognitive Behavioral Stress Management from the patient perspective. Satisfaction measured using the Satisfaction Scale (8 items; 5 = strongly agree, 1 = strongly disagree), which was adapted specifically for this study. A mean satisfaction score will be computed from the 8 items.
Satisfaction (patient perspective 2 of 2) | Week 8
  Assess the satisfaction of telehealth-delivered Cognitive Behavioral Stress Management from the patient perspective using 4 open-ended questions designed specifically for this study. A qualitative summary will be provided based on responses to the open ended questions.

SECONDARY OUTCOMES:
Anxiety symptom improvement | Week 0, 2, 4, 6, 8, 20
  Assess changes in anxiety throughout study using the Generalized Anxiety Disorder 7-item Scale (GAD-7), which asks participants to rate how much they have been bothered by anxiety symptoms over the past 2 weeks (7 items, 0 = not at all, 1= several days, 2= more than half the days 3 = nearly every day). A total score will be created by summing the scores of the 7 items.
Depression symptom improvement | Week 0, 2, 4, 6, 8, 20
  Assess changes in depression throughout study using the Patient Health Questionnaire 9-item Scale (PHQ-9), which asks participants to rate how much they have been bothered by depression symptoms over the past 2 weeks (9 items, 0 = not at all, 1= several days, 2= more than half the days 3 = nearly every day). A total score will be created by summing the scores of the 9 items.

CONTACTS AND LOCATIONS:
Overall Officials: CJ Bathgate, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bathgate CJ, Kilbourn KM, Murphy NH, Wamboldt FS, Holm KE. Pilot RCT of a telehealth intervention to reduce symptoms of depression and anxiety in adults with cystic fibrosis. J Cyst Fibros. 2022 Mar;21(2):332-338. doi: 10.1016/j.jcf.2021.07.012. Epub 2021 Aug 5. PMID 34366282